CLINICAL TRIAL: NCT05604651
Title: Comparison of Mucin Levels at the Ocular Surface of Visual Display Users With and Without Dry Eye Disease
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VDT
Record Dates: First submitted 2022-10-29; First posted 2022-11-03 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-10

CONDITIONS: Dry Eye Disease
Keywords: Dry Eye Disease; Mucin
MeSH Terms: conditions — Dry Eye Syndromes; Medullary cystic kidney disease 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Conjunctival impression cytology samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dry eye disease: Dry eye disease was diagnosed according to the Tear Film and Ocular Surface Society (TFOS) DEWS II criteria: (1) Ocular Surface Disease Index (OSDI) score ≥ 13 and (2) one of these signs; fluorescein tear breakup time (TBUT) <10 sec; abnormal ocular surface staining (>5 corneal spots or > 9 conjunctival spots).
  Interventions: Other: no intervention
- control: The controll group enrolled healthy participants without ocular and systemic diseases.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The study aimed to evaluate 1) if levels of the glycocalyx membrane mucins, including MUC1, MUC4, MUC16 and MUC20, are altered in conjunctival cells of visual display users With and Without Dry Eye Disease, and 2) if mucin levels correlate with dry eye clinical diagnostic data.

DETAILED DESCRIPTION:
The cross-sectional study aimed to evaluate 1) if levels of the glycocalyx membrane mucins, including MUC1, MUC4, MUC16 and MUC20, are altered in conjunctival cells of visual display users With and Without Dry Eye Disease, and 2) if mucin levels correlate with dry eye clinical diagnostic data.

ELIGIBILITY:
Inclusion Criteria:

* Participants who exposed to video display terminals for more than 1 year (at least 5 days per week and 6 hours per day) were enrolled and divided into two groups: (1) VDT users with DED and (2) VDT users without DED. DED was diagnosed according to the Tear Film and Ocular Surface Society (TFOS) DEWS II criteria: (1) Ocular Surface Disease Index (OSDI) score ≥ 13 and (2) one of these signs; fluorescein tear breakup time (TBUT) <10 sec; abnormal ocular surface staining (>5 corneal spots or > 9 conjunctival spots).

Exclusion Criteria:

* a history of contact lens wear or ocular surgery within 2 year of the study visit; a history of previous ocular disease; topical or systemic therapies other than artificial tears within two weeks before recruitment; and inflammatory ocular diseases, ocular surface diseases, glaucoma and systemic diseases with ocular involvement, such as meibomian gland dysfunction, diabetes, and peripheral neuropathy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Video display terminals users with and without dry eye disease.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
mucin expression | immediately after meeting the inclusion and exclusion criteria
  The mRNA expression of mucin was measured by Quantitative real-time PCR, which is a laboratory technique of molecular biology to find out how much of a specific section of DNA there is in a sample.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Qi, PhD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China